CLINICAL TRIAL: NCT03637946
Title: Release of Organic Components of a GIOMER in Non-carious Cervical Lesion Restorations: in Vitro and in Vivo Studies
Brief Title: Release of Organic Components of a GIOMER in Non-carious Cervical Lesion Restorations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government); Fundação de Amparo à Pesquisa do estado de Minas Gerais (Other)
Responsible Party: Principal Investigator, Tassiana Cançado Melo Sá, Principal Investigator, Federal University of Minas Gerais
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FUMinasGerais02; RBR-8m8cf2 (Registry Identifier: Registro Brasileiro de Ensaios Clínicos)
Record Dates: First submitted 2018-08-10; First posted 2018-08-20 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Non-carious Cervical Lesions
Keywords: Resin composite; clinical trial; biocompatibility; cytokines

STUDY DESIGN:
Intervention Model Description: This is a single-center, non-blinded, clinical trial 6 months in duration.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SHOFU Beautifil II LS (Experimental): Experimental: SHOFU Beautifil II LS Restorative system FL-Bond II (self-etching adhesive system)/ Beautifil II (composite restorative)
  Interventions: Other: Device: SHOFU beautifil II LS

INTERVENTIONS:
Other: Device: SHOFU beautifil II LS — Restorative system FL-Bond II (self-etching adhesive system)/ beautifil II (composite restorative) were used following manufacturer's instructions

SUMMARY:
To evaluated the clinical performance of composite resin restorations, considering also the evaluation of release of resin components into saliva and the presence cytokines in gingival fluid. Restorative system FL-Bond II (self-etching adhesive system)/ beautifil II (composite restorative) were use. For in vitro assays, adhesive and resin specimens are being preparing for assessing the monomers degree of conversion (by FTIR), sorption and solubility and release of resinous components in ethanol and Ringer solutions (through a gas chromatography and mass spectroscopy - GC-MS). In the longitudinal clinical study clinical performance of restorations and periodontal response were evaluate.

DETAILED DESCRIPTION:
Release of components of a resin composite system containing pre-reagent vitreal particles: laboratory and patient studies. The objectives of this study was to evaluate physical and chemical properties of a methacrylate-based restorative system regarding to the release of resin components to the storage medium, to evaluate the clinical performance of composite resin restorations, considering also the evaluation of release of resin components into saliva and the presence of cytokines in gingival crevicular fluid. Restorative system FL-Bond II (self-etching adhesive system)/ beautifil II (composite restorative) were use. For in vitro assays, adhesive and resin specimens are being preparing for assessing the monomers degree of conversion (by FTIR), sorption and solubility and release of resinous components in ethanol and Ringer solutions (through a gas chromatography and mass spectroscopy - GC-MS). In the longitudinal clinical study, patients who present a NCCL with restorative need were selecting. Prior to treatment, there will be periodontal evaluation, saliva and gingival crevicular fluid collection (controls). The lesions were restoring with the restorative system. After 10 min,7 days, 1 and 6 months, clinical performance of restorations and periodontal response were evaluate according to the criterion FDI. Additionally, in all of these evaluation periods samples of saliva and crevicular fluid are being collecting. Saliva samples will be analyze by GC-MS to identify the eventual presence of organic components derived from the restoration. The crevicular fluid samples were analyzing using ELISA for identification and quantification of interleukins.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age; Systemically healthy; Non-smoking;
* With good oral hygiene;
* Absent irreversible pulpal alteration;
* With the presence of a non-carious cervical lesion (LCNCs) that needs to be restored. This lesion should be non-carious, non-retentive, with at least 1 mm and up to 3 mm depth, should involve both enamel and dentin of vital teeth without mobility, and present hypersensitivity;
* Presence a natural tooth of the same position of the restored tooth, but in the opposite arch of the same jaw to be considered for the positive control;
* Periodontal parameters : Depth Probing (PS), Visible Plaque Index (IPV), Gingival Index (GI) and Probing Bleed Index (SS). The normal included were: PS = 1 to 3 mm, GI = 0, IPV = score 0 e SS = score 0.

Exclusion Criteria:

* With severe systemic alteration;
* In the use of antibiotics and anti-inflammatories in the last three months;
* With periodontium with periodontal parameters different from those established in the inclusion criteria.
* Individuals with clinical signs of parafunctional habits;
* Smoking;
* Individuals who have performed other restorations in the last 12 months;
* Pregnant women and infants;
* Periodontal sites that presented bleeding during crevicular fluid collection or sites that prevent proper collection of clinical parameters.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
FDI criteria | Up to 6 months
  The evaluation of the quality of the restoration will be evaluated using the FDI criteria and will be performed by two trained examiners at baseline and follow-up visits.The criteria has score given for each property with range from 1 to 5. Clinical assessments (Esthetic properties:surface brightness, surface and marginal color, color and translucency and anatomical form, Functional properties: marginal adaptation, fracture of material and retention, and Biological Properties: postoperative hypersensitivity, recurrence of caries, tooth integrity and adjacent mucosa)

SECONDARY OUTCOMES:
Clinical parameters: visible plaque index (IPV) | T1:One week before of starting treatment;T2: After 10 minutes of starting treatment;T3: After 1 week of starting treatment;T4: After 30 days of starting treatment;T5:After 6 months
  registered presence (score 1) or absence (score 0) of bacterial plaque without the use of probe, after drying the dental surface with compressed air.
Clinical parameters: probing depth (PS) | T1:One week before of starting treatment;T2: After 10 minutes of starting treatment;T3: After 1 week of starting treatment;T4: After 30 days of starting treatment;T5:After 6 months;
  distance from the gingival margin to the fundus of the gingival sulcus or periodontal pocket, which will be measured by means of manual circumferential probing and measured on all the faces of the restored teeth and control;
Clinical parameters: probing bleeding (SS) | T1:One week before of starting treatment;T2: After 10 minutes of starting treatment;T3: After 1 week of starting treatment;T4: After 30 days of starting treatment;T5:After 6 months
  Bleeding to the Survey (SS): evaluated at the moment of PS measurement or until 30 to 60 seconds after the introduction of the probe with dichotomic values by presence (score 1) or absence (score 0)
Clinical parameters: gingival index (GI) | T1:One week before of starting treatment;T2: After 10 minutes of starting treatment;T3: After 1 week of starting treatment;T4: After 30 days of starting treatment;T5:After 6 months
  evaluates the existence and severity of gingival lesions on a scale ranging from 0 to 3, where: 0: normal;
  1. mild inflammation with color change, mild edema, no bleeding at probing;
  2. moderate inflammation with red, shiny, swollen gingival tissue and presence of bleeding on probing;
  3. severe inflammation, with great increase of color and edema, ulceration and tendency to spontaneous bleeding.

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University Of Minas Gerais, Belo Horizonte, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No